CLINICAL TRIAL: NCT00636376
Title: Effect of Head Elevation on Intracranial Pressure and Cerebral Venous Outflow in Children
Brief Title: Effects of Head Elevation on Intracranial Pressure in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Jimmy Huh, MD, The Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2002-1-2721
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Head Injury
Keywords: elevated intracranial pressure; inadequate cerebral perfusion; secondary brain damage
MeSH Terms: conditions — Craniocerebral Trauma; Intracranial Hypertension | interventions — Intracranial Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Single arm--no randomization. All subjects enrolled will have vitals collected and three ultrasounds at different levels of head of the bed elevations.
  Interventions: Procedure: Place HOB in alternate positions from 0-50 degrees.

INTERVENTIONS:
Procedure: Place HOB in alternate positions from 0-50 degrees. — Patients will receive an US while the HOB(Elevation of the head of bed) is 30 degrees(baseline) then they will increase the angle to 40 degrees, then 50 degrees. Another US will be done then in 20, 10, and o degree angles. Then another US will be done
  Other Names: Intracranial Pressure; Cerebral Venous Outflow; Head Elevation; Traumatic brain injury; Head injury

SUMMARY:
Head injury is the most common cause of mortality and acquired disability in childhood. It is common to elevate the head of patients at risk for increased intracranial pressure, although it is not clear if it is always beneficial. Every severe pediatric traumatic brain injured patient will have an optimal head position that prevents rising pressure in the brain.

DETAILED DESCRIPTION:
Head injury is the most common cause of mortality and acquired disability on childhood. Management of children at risk for intracranial hypertension is both complex and increasingly controversial. Also, effect of head position on intracranial pressure, cerebral perfusion pressure, adn cerebral venous outflow in the pediatric population has not been studied. We will examine the effect of head positioning on ICP, CPP, and cerebral venous outflow in pediatric patients at risk for intracranial hypertension. The hypothesis is that ICP will be reduced with improvement in cerebral venous outflow by each patient having their own optimal head position.

ELIGIBILITY:
Inclusion Criteria:

* Neonates, children, and adolescents
* Intracranial pressure monitor in place

Exclusion Criteria:

* Severe multiorgan system failure
* Hemodynamic instability sufficient to preclude changes in head position

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2002-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
ICP will be reduced with improvement in cerebral venous outflow which is dependent on intravascular volume status and intrathoracic pressure and each will have their own optimal head position. | As long as ICP is being monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Huh, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States